CLINICAL TRIAL: NCT00670189
Title: A Phase 1 Multiple Ascending Dose Study of BMS-833923 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 Study of BMS-833923 (XL139) in Subjects With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA194-002
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Hedgehog Pathway; Smoothened; Basal Cell Carcinoma (BCC); Basal Cell Nevoid Syndrome (BCNS)
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — BMS-833923

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-833923 (Experimental)
  Interventions: Drug: BMS-833923 (XL139)

INTERVENTIONS:
Drug: BMS-833923 (XL139) — Capsules, Oral, 30 mg starting; dose escalation, Once daily, 37 days; additional days if receiving benefit

SUMMARY:
The purpose of this study is to determine the safety of BMS-833923 (XL139) in patients with advanced or metastatic cancers and determine the recommended phase 2 dose range and schedule

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Advanced or metastatic cancer (excluding cancer in the blood) or uncontrolled basal cell nevoid syndrome or sporadic basal cell carcinoma
* Primary or metastatic tumor site accessible for biopsy
* Ability to swallow capsules
* Subjects with histologically confirmed, advanced stage IIIB or stage IV non-small cell lung cancer (NSCLC) with a primary histology of squamous carcinoma who have received prior systemic therapy for advanced NSCLC will be enrolled in Part 3

Exclusion Criteria:

* Uncontrolled brain metastasis
* Significant cardiovascular disease
* Inadequate blood counts
* Inadequate liver, kidney or lung function
* Gastrointestinal disease within last 3 months
* Infection with Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C or exposure to attenuated active immunizations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-07; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Use National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) to establish the maximum tolerated dose, a recommended Phase 2 dose range and schedule, and safety profile of BMS-833923 | On average a minimum of 60 days up to 3 years
  Use NCI CTCAE to monitor safety assessments including physical findings, laboratory tests, and radiographic assessments to establish the maximum tolerated dose and recommended Phase 2 dose range and schedule of BMS-833923

SECONDARY OUTCOMES:
Pharmacokinetic parameters of BMS-833923 (XL139) following a single-dose and during daily dosing: Maximum observed plasma concentration (Cmax) | Study day 1-7, 36
Pharmacokinetic parameters of BMS-833923 (XL139) following a single-dose and during daily dosing: Time of maximum observed plasma concentration (Tmax) | Study day 1-7, 36
Pharmacokinetic parameters of BMS-833923 (XL139) following a single-dose: Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-t)] of BMS-833923 (XL139) | Study day 1-7
Pharmacokinetic parameters of BMS-833923 (XL139) following a single-dose: Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-833923 (XL139) | Study day 1-7
Pharmacokinetic parameters of BMS-833923 (XL139) following a single-dose: Plasma half-life (T-HALF) of BMS-833923 (XL139) | Study day 1-7
Pharmacokinetic parameters of BMS-833923 (XL139) during daily dosing: Minimum observed plasma concentration (Cmin) of BMS-833923 (XL139) | Study day 1, 8, 15, 22, 29, 36, 64, and 92
Pharmacokinetic parameters of BMS-833923 (XL139) during daily dosing: Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-833923 (XL139) | Study day 36
To assess the pharmacodynamic effects of BMS-833923 (XL139) on Hedgehog (HH) pathway activation in skin by evaluation of biomarkers such as, but not limited to GLI-1 protein or mRNA expression using immunohistochemistry (IHC) or RT-PCR in a skin biopsies | At screening (baseline) and between days 22 and 36 of treatment
  glioma-associated oncogene family of transcription factors (GLI)
To assess the pharmacodynamic effects of BMS-833923 (XL139) on HH pathway activation in subjects' tumors by evaluation of protein and mRNA of biomarkers such as, but not limited to GLI-1, in pre- and during-treatment tumor samples | At screening (baseline) and between days 22 and 36 of treatment. At screening only for NSCLC patients
  glioma-associated oncogene family of transcription factors (GLI)
To describe any preliminary evidence of anti-tumor activity of BMS-833923 (XL139) | Every 8 weeks until disease progression
  Tumor assessments by computed tomography (CT)
Safety profile of multiple doses of BMS-833923 | Adverse event reports: On average a minimum of 60 days up to 3 years
  Medical review of adverse event reports
Safety profile of multiple doses of BMS-833923 | Conducted at least on days 1, 8, 15, 22 and 36 of the first 36-day cycle and then monthly or biweekly for the first 6 months, then monthly
  The results of vital sign measurements, electrocardiogram (ECGs), pulmonary function tests, multigated radionuclide angiography (MUGA) or echocardiograms, physical examinations, and clinical laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (2):
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Southwest Texas Addiction Research And Tech (Start) Center, San Antonio, Texas
- Local Institution, Toronto, Ontario, Canada

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx